CLINICAL TRIAL: NCT00739232
Title: Single Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HSD-016 Administered Orally to Healthy Subjects
Brief Title: Single Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HSD-016
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3248A1-1000
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
Keywords: Safety and tolerability of HSD-016
MeSH Terms: interventions — (R)-1,1,1-trifluoro-2-(3-((R)-4-(4-fluoro-2-(trifluoromethyl)phenyl)-2-methylpiperazin-1-ylsulfonyl)phenyl)propan-2-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Active
  Interventions: Drug: HSD-016
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: HSD-016
  Arms: Active
Other: placebo
  Arms: Placebo

SUMMARY:
This is a single ascending dose study of HSD-016 to provide the initial assessment of the safety, tolerability, how the drug is absorbed and eliminated, and its effect on the body.

ELIGIBILITY:
Inclusion:

1. Men or women of nonchildbearing potential aged 18 to 50 years inclusive at screening.
2. Healthy as determined by the investigator on the basis of screening evaluations.
3. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history.

Exclusion:

1. No presence or history of any disorder that may prevent the successful completion of the study.
2. No history of drug abuse within 1 year.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 3 months

SECONDARY OUTCOMES:
Profiles of Drug Concentrations | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Overland Park, Kansas, United States